CLINICAL TRIAL: NCT05052723
Title: Phase II Clinical Trial Evaluating Cabozantinib and Pembrolizumab in Metastatic Pancreatic Cancer
Brief Title: Cabozantinib and Pembrolizumab in Metastatic Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Kim (Other)
Collaborators: Exelixis (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Joseph Kim, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21-GI-117
Record Dates: First submitted 2021-09-12; First posted 2021-09-22 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
Keywords: Adenocarcinoma; Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — cabozantinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib and pembrolizumab (Experimental)
  Interventions: Drug: Cabozantinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib (XL184) is a potent inhibitor of multiple receptor tyrosine kinases (RTKs) known to play important roles in tumor cell proliferation and/or tumor neovascularization.
Drug: Pembrolizumab — Pembrolizumab is a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD-1) receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2).

SUMMARY:
This study aims to evaluate cabozantinib and pembrolizumab for the treatment of metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatic ductal adenocarcinoma
* Evidence of progression or intolerance to previous standard of care pancreatic cancer systemic or locoregional therapies
* Patients must have adequate organ function

Exclusion Criteria:

* Chemotherapy or other locoregional anti-tumoral therapies performed within 28 days of study treatment initiation
* Received palliative radiation therapy within 2 weeks or any other radiation therapy within 4 weeks of start of study intervention
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation
* Has a diagnosis of immunodeficiency (autoimmune disease) or is receiving chronic systemic steroid therapy
* Clinically significant cardiovascular disease
* Uncontrolled hypertension
* Inability to swallow tablets

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josepoh Kim, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald HG, Cassim EB, Harper MM, Burke EE, Marcinkowski EF, Cavnar MJ, Pandalai PK, Kim J. The Development of Investigator-Initiated Clinical Trials in Surgical Oncology. Surg Oncol Clin N Am. 2023 Jan;32(1):13-25. doi: 10.1016/j.soc.2022.07.003. Epub 2022 Nov 3. PMID 36410913

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib and pembrolizumab
Started | 21
Completed | 2
Not Completed | 19
Not completed — Death | 19

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib and Pembrolizumab
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progress-free survival in participants, defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever comes first.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and pembrolizumab
Number analyzed (Participants) | 21
Participants | 2

2. Secondary Outcome: Number of Participants With Response to Therapy
Description: The proportion of participants with overall response to therapy via imaging; Overall Response Rate (%) = (Number of patients achieving Complete responses + Number of patients achieving partial responses / Total Number of patients) × 100
Time Frame: 1 year
Population: Number of participants with complete or partial response reported
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and pembrolizumab
Number analyzed (Participants) | 21
Participants | 1

3. Secondary Outcome: Number of Participants With Complete Response
Description: The proportion of participants with a complete response to therapy
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and pembrolizumab
Number analyzed (Participants) | 21
Participants | 0

4. Secondary Outcome: Number of Participants With Partial Response
Description: The proportion of participants with a partial response to therapy
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and pembrolizumab
Number analyzed (Participants) | 21
Participants | 1

5. Secondary Outcome: Overall Participant Survival Rate
Description: Overall survival rate participants
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and pembrolizumab
Number analyzed (Participants) | 21
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 year
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting
Arm/Group | Cabozantinib and pembrolizumab
All-Cause Mortality (participants affected / at risk) | 19/21
Serious Adverse Events (participants affected / at risk) | 13/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib and pembrolizumab (N=21)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Disease Progression (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Endocarditis Infective (Infections and infestations) | 1 (1)
Other (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (4)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Stroke (Nervous system disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (4)
Dysuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib and pembrolizumab (N=21)
Anemia (Blood and lymphatic system disorders) | 6 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (3)
Mitral valve disease (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Ascites (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (4)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 11 (18)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Other (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 11 (15)
Vomiting (Gastrointestinal disorders) | 7 (8)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 5 (6)
Fatigue (General disorders) | 14 (21)
Fever (General disorders) | 2 (3)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 4 (4)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Other (Infections and infestations) | 1 (1)
Infective myositis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (16)
Alkaline phosphatase increased (Investigations) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 10 (16)
Blood bilirubin increased (Investigations) | 1 (1)
Cardiac troponin I increased (Investigations) | 2 (2)
Cardiac troponin T increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 2 (5)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (9)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 6 (7)
Thyroid stimulating hormone increased (Investigations) | 3 (3)
Urine output decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 3 (6)
White blood cell decreased (Investigations) | 2 (2)
Metabolism and nutrition disorders (Investigations) | 14 (83)
Alkalosis (Investigations) | 1 (1)
Anorexia (Investigations) | 10 (11)
Dehydration (Investigations) | 3 (4)
Hyperglycemia (Investigations) | 5 (10)
Hyperkalemia (Investigations) | 3 (9)
Hypermagnesemia (Investigations) | 1 (1)
Hypernatremia (Investigations) | 1 (1)
Hypoalbuminemia (Investigations) | 8 (9)
Hypocalcemia (Investigations) | 11 (18)
Hypokalemia (Investigations) | 4 (4)
Hypomagnesemia (Investigations) | 3 (3)
Hyponatremia (Investigations) | 7 (11)
Hypophosphatemia (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (7)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (8)
Dysarthria (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (4)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Lethargy (Nervous system disorders) | 1 (1)
Muscle weakness right-sided (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Psychiatric disorders (Nervous system disorders) | 5 (5)
Anxiety (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 2 (2)
Insomnia (Nervous system disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Glucosuria (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Other (Skin and subcutaneous tissue disorders) | 1 (3)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 8 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT05052723/Prot_SAP_000.pdf